CLINICAL TRIAL: NCT04802096
Title: Effects of Inspiratory Muscle Training in Addition to Pulmonary Rehabilitation in Patients With COPD Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202012102RINC
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Exacerbation Copd

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training combined pulmonary rehabilitation (Experimental)
  Interventions: Other: inspiratory muscle training; Other: pulmonary rehabilitation
- Sham inspiratory muscle training combined pulmonary rehabilitation (Sham Comparator)
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: inspiratory muscle training — Intensity of inspiratory muscle training will be set at 30% of maximal inspiratory pressure. Subjects in intervention experimental group will perform 15 breaths per set, 6 sets per day on daily basis. The intervention will be last for 8 weeks.
  Arms: Inspiratory muscle training combined pulmonary rehabilitation
Other: pulmonary rehabilitation — Pulmonary rehabilitation consists of aerobic exercise training, strength training, and education related to airway clearance and drug utilization. All of subjects will receive 8-week pulmonary rehabilitation.

SUMMARY:
Inspiratory muscle weakness, limited functional exercise capacity and worse quality of life have been shown in patients with exacerbation of chronic obstructive pulmonary disease (COPD). Recommendations from clinical practice guideline state that promoting pulmonary rehabilitation after exacerbation can improve the conditions above. Inspiratory muscle training (IMT) has been proven to enhance inspiratory muscle strength and endurance in patient with stable COPD. However, there is less research on whether IMT in addition to pulmonary rehabilitation after exacerbation can benefit inspiratory muscle function, functional exercise capacity and quality of life in patients with COPD. The purpose of this study is to examine the effects of IMT in addition to pulmonary rehabilitation on respiratory muscle function, functional exercise capacity and quality of life in patients with exacerbation of chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years old
* diagnosed as exacerbation of COPD
* maximal inspiratory pressure (MIP) < 80 cmH2O

Exclusion Criteria:

* any clinical diagnosis that will influence the measurement, including any history of neuromyopathy
* angina, acute myocardial infarction in the previous one month
* pregnancy
* participated in inspiratory muscle training program in the previous three months
* any psychiatric or cognitive disorders, for example: Mini-Mental State Examination (MMSE) < 24, that will disturb the communication and cooperation of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Diaphragm muscle activation | 10 minutes
  The surface electromyography (EMG) signal was analyzed in the time domain, calculating root mean square (RMS) amplitude with a time constant of 30 mini seconds. A 1.5 seconds window of diaphragm muscle signals at peak pressure during maximal inspiratory pressure test were obtained and calculated as maximal effort. Diaphragm activation were calculated using mean RMS values of each threshold loaded breathing test, and then normalized to maximal effort (%EMGDia).
Sternocleidomastoid muscle activation | 10 minutes
  The surface electromyography (EMG) signal was analyzed in the time domain, calculating root mean square (RMS) amplitude with a time constant of 30 mini seconds. A 1.5 seconds window of SCM muscle signals at peak pressure during maximal inspiratory pressure test were obtained and calculated as maximal effort. SCM activation were calculated using mean RMS values of each threshold loaded breathing test, and then normalized to maximal effort (%EMGSCM).

SECONDARY OUTCOMES:
The mean median frequency of diaphragm and sternocleidomastoid muscle | 10 minutes
  The power spectrum is divided into two equal areas of the frequency value by median frequency to exam muscle fatigue.
Functional exercise capacity | Considering time of test and recovery, it will be expected to take totally 10 minutes.
  Six-minute walking test will be performed to evaluate functional exercise capacity.
Quality of life evaluation | 10 minutes
  St. George's Respiratory Questionnaire and COPD assessment test will be used to evaluate quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, PhD, Study Chair — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy of National Taiwan University, Taipei, Zhongzheng Dist, Taiwan

REFERENCES:
- [Derived] Huang WY, Lee CT, Chien JY, Hsu M, Wang LY. Effects of Inspiratory Muscle Training in Patients With Chronic Obstructive Pulmonary Disease Exacerbations: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 May 1;104(5):458-464. doi: 10.1097/PHM.0000000000002654. Epub 2024 Nov 11. PMID 39774113